CLINICAL TRIAL: NCT03957590
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Tislelizumab (BGB-A317) Versus Placebo in Combination With Concurrent Chemoradiotherapy in Patients With Localized Esophageal Squamous Cell Carcinoma
Brief Title: A Study to Investigate Tislelizumab (BGB-A317) Versus Placebo in Combination With Concurrent Chemoradiotherapy in Participants With Localized Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGB-A317-311; CTR20190198 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab + chemoradiotherapy (Experimental): Tislelizumab once every 3-week cycle (Q3W) + paclitaxel on Day 1 of every cycle, for a total of 2 cycles + cisplatin on Day 1 to 3 of every cycle (3 weeks), for a total of 2 cycles + Radiotherapy
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy
- Placebo combined + chemoradiotherapy (Placebo Comparator): Placebo once every 3-week cycle (Q3W) + paclitaxel on Day 1 of every cycle, for a total of 2 cycles + cisplatin on Day 1 to 3 of every cycle (3 weeks), for a total of 2 cycles + Radiotherapy
  Interventions: Drug: Placebo; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Administrated at dose of 200 mg intravenously (IV)
  Other Names: BGB-A317
  Arms: Tislelizumab + chemoradiotherapy
Drug: Placebo — Placebo to match tislelizumab
  Arms: Placebo combined + chemoradiotherapy
Drug: Paclitaxel — Administered as 135 mg/m² IV injection
Drug: Cisplatin — Administered as 25 mg/m² IV injection
Radiation: Radiotherapy — Administered at a total dose of 50.4 Gy in 28 fractions

SUMMARY:
This is a phase 3, randomized, double-blind, placebo-controlled study to compare the efficacy and safety of BGB-A317 versus placebo with chemoradiotherapy in participants with Localized Esophageal Squamous Cell Carcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 75 years on the day of signing the informed consent form
* Histologically confirmed diagnosis of localized ESCC
* Measurable and/or non-measurable disease defined per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Adequate organ function

Key Exclusion Criteria:

* Indicators of severe malnutrition
* Clinically uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention within 2 weeks prior to randomization
* Known to be intolerable or resistant to treatment with the protocol-specified chemotherapy
* Received prior radiotherapy or therapies targeting PD-1, PD-L1, PD-L2 or other immune-oncology therapies
* Active autoimmune diseases or history of autoimmune diseases that may relapse

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization up to 4 years, approximately
  PFS is- defined as the time from randomization to the first documented disease progression, as determined by the Blinded Independent Review Committee (BIRC) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization up to 4 years, approximately
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Change from baseline in European Quality of Life-Core 30 Questionnaire index (EORTC QLQ-C30) | Baseline to end of treatment ~2 years
  The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 =Not at all (best) to 4 =Very Much (worst) and 2 questions answered on a 7-point scale where 1 =Very poor (worst) to 7 =Excellent (best).
Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire esophageal cancer module (EORTC QLQ-OES18) | Up to 2 years, approximately
  Total of 18 questions to assess your symptoms or problems during the past week, each assessed on a scale from 1 (not at all) to 4 (very much). with the range from minimum scores 1 as better outcome and maximum 4 as worst outcomes. Symptoms includes whether any difficulty to eating solids, liquidized or softs food, drinking, or not， whether it is difficult to or swallowing, trouble eating or enjoying meals, pain when eating, dry mouth, food tasting differently, trouble talking, ， whether the sense of smell and conversation are normal or not， whether have Symptoms include cough, indigestion or heartburn, acid reflux and pain or not in the chest or stomach.
Overall response rate (ORR) | From date of randomization up to 4 years, approximately
  ORR is defined as the percentage of participants who had complete response (CR) or partial response (PR) as assessed by BIRC per RECIST v1.1
Duration of response (DOR) | From first determination of an objective response up to 4 years, approximately
  DOR is defined as the time from the first occurrence of a documented objective response to the time of relapse, as determined by the BIRC per RECIST v1.1, or death from any cause, whichever occurs first
Number of Participants with treatment-emergent adverse events (TEAEs) | Up to 2 years, approximately
  Adverse events will be graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Weihu Wang, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Zefen Xiao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (33):
- China (33):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospitalschool of Clinical Medicine of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Jieyang Peoples Hospital (Jieyang Affiliated Hospital, Sun Yat Sen University ), Jieyang, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Inner Mongolia Autonomous Region Cancer Hospital, Hohhot, Inner Mongolia
  - Changzhou Tumor(Fourth Peoples)Hospital, Changzhou, Jiangsu
  - The First Peoples Hospital of Lianyungang, Lianyungang, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu Peoples Hospital, Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Derived] Yu R, Wang W, Li T, Li J, Zhao K, Wang W, Liang L, Wu H, Ai T, Huang W, Li L, Yu W, Wei C, Wang Y, Shen W, Xiao Z. RATIONALE 311: tislelizumab plus concurrent chemoradiotherapy for localized esophageal squamous cell carcinoma. Future Oncol. 2021 Nov;17(31):4081-4089. doi: 10.2217/fon-2021-0632. Epub 2021 Jul 16. PMID 34269067